CLINICAL TRIAL: NCT01733693
Title: Neurocognitive Effects of Opiate Agonist Treatment
Acronym: NEO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Montefiore Medical Center (Other); Fordham University (Other)
Responsible Party: Principal Investigator, Julia H. Arnsten, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-433; 1R01DA032552-01A1 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-27 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Opioid-Related Disorders; HIV; HIV Infections
Keywords: Buprenorphine; Methadone; Cognition
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections | interventions — Buprenorphine; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine (Experimental): Oral sublingual tablet, 8-32 mg per day, administered daily for duration of 4 months
  Interventions: Drug: Buprenorphine
- Methadone (Active Comparator): Oral sublingual tablet, 60-100 mg per day, administered daily for duration of 4 months
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Buprenorphine — Study participants will be randomly assigned 1:1 to buprenorphine (experimental/intervention) or methadone (active comparator). We will stratify by HIV status to ensure an equal number of HIV-infected participants in each group.
  Other Names: Buprenorphine HCl
  Arms: Buprenorphine
Drug: Methadone — Study participants will be randomly assigned 1:1 to buprenorphine (experimental/intervention) or methadone (active comparator). We will stratify by HIV status to ensure an equal number of HIV-infected participants in each group.
  Other Names: Methadone Hydrochloride
  Arms: Methadone

SUMMARY:
The purpose of this study is to (1) compare the effects of buprenorphine and methadone, two types of opioid addiction treatment, on the ability to think and reason among people addicted to opiates, and who are either HIV negative or HIV positive; and (2) investigate whether HIV infection changes the way opioid treatment affects the ability to think and reason. The investigators hypothesize that there will be (1) significant improvement in thinking and reasoning ability after starting buprenorphine treatment compared to methadone treatment, among participants with and without HIV at 2 and 4 months compared to baseline; and (2) HIV positive participants will demonstrate significant improvement in thinking and reasoning ability at 2 and 4 months compared to baseline, but that their thinking and reasoning ability will still be lower than HIV negative participants.

DETAILED DESCRIPTION:
After randomization, each medication will be prescribed and administered by one of these experienced clinicians, according to well- established national protocols. Participants will be randomized in a 1:1 ratio in variable size blocks of 4-8 via central, computer-generated randomization. Given the relatively small sample size, we will randomize in blocks to ensure comparison groups of approximately equal size. Because medication type will not be blinded, we will vary block size to prevent anticipation of treatment arm assignment. We will also stratify randomization by HIV status to ensure equal numbers of HIV-infected persons in each arm.

INTERVENTION DOSE. Doses of buprenorphine and methadone will be adjusted within pre-specified ranges to ensure that comparisons between the two treatments are based on individually optimized doses.

Buprenorphine (we will use the buprenorphine/naloxone combination exclusively) will be administered at a dose of 8 to 32 mg per day, though we expect most subjects not to exceed 24 mg per day. These doses approximate methadone doses of 60 to 100 mg daily, which are in the upper range of doses generally used in clinical practice, but are well-known to be most efficacious and are also most prevalent in DoSA. Since study clinicians will be experienced substance abuse treatment providers, some flexibility will be allowed within these parameters. Both buprenorphine and methadone will be administered daily as oral medications.

The study will have two phases: induction/stabilization (weeks 1 - 3) and maintenance (weeks 4 - 24).

During dose induction/stabilization, subjects will attend daily visits (Sx/week) with a study clinician and receive gradually increasing doses of medication (see below). The first week of induction/stabilization will be considered a run-in period; at the conclusion of this week participants will complete enrollment in the trial and also complete their first NP research visit. The purpose of the run-in period is to ensure that we enroll persons who are able to comply with all trial requirements.

MAINTENANCE PHASE. The maintenance stage of opioid pharmacotherapy begins when a patient is responding optimally to medication treatment and routine dosage adjustments are no longer needed. Patients at this stage have stopped abusing opioids and many remain on the same dosage of treatment medication for many months, whereas others require frequent or occasional adjustments. During maintenance (starting on day 22, week 4),subjects in both arms will attend the clinic three times per week, on Monday, Wednesday, and Friday, and will receive bottles of medication to take home for the other four days of the week. Subjects will receive increases in their doses starting in week 4 if they meet pre-established criteria, up to 100 mg of methadone, and up to 32 mg of buprenorphine.

Our proposed research plan includes two follow-up visits, three and six months after the baseline visit. We anticipate that subjects will still be in the maintenance phase at the time of both these visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 68
* English or Spanish speaking
* Documentation of HIV Status
* Opioid-dependent without having received medication treatment for opioid dependence within the previous 90 days
* Negative pregnancy test, for women
* No "street" use of methadone or buprenorphine
* Willing to participate in all study components
* Able to provide informed consent
* Education > 6 years
* Not acutely intoxicated

Exclusion Criteria:

* Serious or unstable medical disease: liver disease (AST or ALT ≥ 3x ULN, elevated PT/INR, albumin <3.0 g/dl or evidence of decompensated cirrhosis);
* Severe cardiovascular disease (MI, PTCA, unstable angina, CABG, and/or serious arrhythmia in the previous 6 months);
* COPD (requiring supplemental oxygen or hospitalization in past 6 months);
* End stage renal disease or creatinine clearance <30 mL/min
* Neurological disease: head injury with LOC>24 hour, previous penetrating skull wound, focal brain lesion, history of neurosurgery, seizure disorder (not ETOH-related), non-HIV CNS opportunistic infection
* Psychiatric disorders (schizophrenia or bipolar)
* Benzodiazepine or alcohol dependence
* Chronic pain conditions requiring opioid analgesics

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Global Neurocognitive Function | 2 and 4 months
  Metrics:
  A Global Deficit Score (GDS) is computed by adding deficit ratings of the component test measures, and dividing by total number of measures. (Please see list of component test measures under the Domain-Specific Neurocognitive Function outcome).
Domain-Specific Neurocognitive Function (i.e. in the domains of executive functioning, learning, memory, attention/working memory, processing speed, motor, and verbal functioning). | 2 and 4 months
  Metrics:
  Domain Deficit Scores (DDS) are created for each of the 7 cognitive ability domains. Deficit Scores can be analyzed as dichotomous variables to classify individual subjects as impaired or normal, or continuously.
  Executive Functioning -- Wisconsin Card Sorting Task-64 Item Version; Trail Making Test (Part B)
  Learning -- Hopkins Verbal Learning Test-Revised (Total Recall); Brief Visuospatial Memory Test-Revised (Total Recall)
  Memory -- Hopkins Verbal Learning Test (Delayed Recall Trial); Brief Visuospatial Memory Test-Revised (Delayed Recall Trial)
  Attention/Working Memory -- WAIS-III Letter Number Sequencing; PASAT Total Correct
  Processing Speed -- WAIS-III Digit Symbol; WAIS-III Symbol Search; Trail Making Test (Part A)
  Motor -- Grooved Pegboard Time (dominant hand); Grooved Pegboard Time (non-dominant hand)]
  Verbal Functioning -- Controlled Oral Word Association Test (F-A-S); Semantic (Animal) Fluency

CONTACTS AND LOCATIONS:
Overall Officials: Julia Arnsten, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Fordham University, The Bronx, New York
  - Albert Einstein College of Medicine of Yeshiva University, The Bronx, New York

REFERENCES:
- [Derived] Scott TM, Arnsten J, Olsen JP, Arias F, Cunningham CO, Rivera Mindt M. Neurocognitive, psychiatric, and substance use characteristics in a diverse sample of persons with OUD who are starting methadone or buprenorphine/naloxone in opioid treatment programs. Addict Sci Clin Pract. 2021 Oct 24;16(1):64. doi: 10.1186/s13722-021-00272-4. PMID 34689841